CLINICAL TRIAL: NCT04269070
Title: WorkWell: A Pre-clinical Pilot Study of Increased Standing and Light-intensity Physical Activity in Prediabetic Sedentary Office Workers
Brief Title: WorkWell: Work-based Activity and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00010172
Record Dates: First submitted 2020-01-03; First posted 2020-02-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes; Obesity
Keywords: sedentary; prediabetes; lifestyle modification; cardiometabolic health
MeSH Terms: conditions — Prediabetic State; Obesity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This is a crossover trial where study participants will experience two conditions following a baseline usua behavior conditions. All study participants will experience each of the conditions: a standing condition, and a light intensity physical activity (LPA) intervention.
Who Masked: Outcomes Assessor
Masking Description: Flow-mediated dilation outcome: Images that are obtained will be analyzed by a blinded researcher using a previously validated, edge-detection software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move, Stand (Active Comparator): Usual behavior condition, followed by the standing condition, followed by the LPA condition.
  Interventions: Behavioral: Standing condition; Behavioral: Light physical activity (LPA) condition; Behavioral: Usual behavior condition
- Stand, Move (Active Comparator): Usual behavior condition, followed by the LPA condition, followed by the standing condition.
  Interventions: Behavioral: Standing condition; Behavioral: Light physical activity (LPA) condition; Behavioral: Usual behavior condition

INTERVENTIONS:
Behavioral: Standing condition — Participants will be asked to stand an additional 6 minutes per hour above their median standing time from the observed time in the usual behavior condition.
Behavioral: Light physical activity (LPA) condition — Participants will be asked to perform 6 additional minutes per hour above their median LPA time from the observed time in the usual behavior condition.
Behavioral: Usual behavior condition — Participants will be asked to perform their normal work activities in their normal work environment for one week. There will be no modifications to their work environment or instructions given of what activities to partake in. This period will be used to understand their normal standing and LPA behaviors to determine the personalized changes to their standing and LPA behaviors in the other conditions.

SUMMARY:
This study will test whether a range of pre-clinical cardiometabolic biomarkers can be improved via regular intervals of standing and light-intensity physical activity in real-world office environments.

DETAILED DESCRIPTION:
This pilot study is being conducted to determine whether a range of pre-clinical cardiometabolic biomarkers (measured via gut microbiome, blood draw) can be improved via regular intervals of standing and light-intensity physical activity (i.e., leisurely walking) in real-world office environments. This trial is meant to generate pilot data which will lead to additional clinical trials.

Primary Hypothesis: Increasing both standing and light-intensity physical activity will improve biomarkers of metabolic function, as measured by blood metabolites and differential abundance of gut microbiome composition, compared to a control condition of normal workplace behavior.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age 18 yrs and older
* Holds a job where primary work activities are done seated
* Has the space and ability to use a sit-to-stand workstation in their primary workspace
* Works in an office setting or remotely for ≥ 4 days per week
* Have a BMI ≥ 25.0 (≥23.0 for individuals of Asian descent)

Exclusion Criteria:

* Currently taking diabetes medication
* Taking any of the following medications or treatments:

  * Medication to control high blood pressure
  * Medication to treat high glucose
  * Blood thinners
  * Hormone replacement therapy (in the past 12 months)
  * Corticosteroids
  * High dose statins (Dr. Reaven, MD to adjudicate eligibility based on dosage)
  * 2nd generation antipsychotics
* Current or previous foot or lower limb injuries
* Current use of sit-stand workstation
* Current smoker
* Neuromuscular or cardiovascular disorders or other serious active medical issues, including deep vein thrombosis or respiratory issues
* Has a physical impairment or musculoskeletal condition that will prevent the subject from standing or light-intensity walking for a maximum of 30 minutes
* Has been advised to avoid prolonged periods of sitting or standing by a physician or other healthcare provider
* History of inflammatory bowel or intestinal malabsorption conditions
* Use of prebiotics, probiotics or antibiotics in the last 3 months
* Serious food allergies or restrictions
* Participants who will be travelling 3 or more days out of their typical week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in 2-hour postprandial area-under-the-curve blood glucose at 2 weeks | 2 weeks
  Participants will be asked to wear the Abbott Freestyle Libre continuous glucose monitor during the usual behavior condition (week 1) and both experimental conditions (weeks 2-3 and weeks 5-6). Research staff will insert the CGM sensor at the screening and study visits. The training for this insertion will be conducted by a registered research nurse. The CGM sensors have been designed and tested to be worn continuously for up to 14 days. Sensors will be placed and removed by trained research staff at appropriate time-points throughout the study. Postprandial period will follow a standardize lunch meal. Area-under-the-curve calculations will be based on 2 hours following delivery of this lunch meal.

SECONDARY OUTCOMES:
Change in baseline workplace standing time at 2 weeks | 2 weeks
  Participants will be asked to wear an activPAL accelerometer throughout the entire intervention period. Data from the devices will be downloaded at each study visit. The activPAL device is worn on the right thigh and is equipped with low energy Bluetooth and will communicate wirelessly with the provided smartphone application to provide feedback to the participant and compliance with the protocol. Workplace time will be assessed by a self-report log and activPAL time will be extracted based on these reports.
Change in baseline workplace stepping time at 2 weeks | 2 weeks
  Participants will be asked to wear an activPAL accelerometer throughout the entire intervention period. Data from the devices will be downloaded at each study visit. The activPAL device is worn on the right thigh and is equipped with low energy Bluetooth and will communicate wirelessly with the provided smartphone application to provide feedback to the participant and compliance with the protocol. Workplace time will be assessed by a self-report log and activPAL time will be extracted based on these reports.

OTHER OUTCOMES:
Treatment acceptability/satisfaction | 2 weeks
  Intervention acceptability questionnaire at the end of each condition will elicit each participant's perceived acceptability of the intervention.
Change in fasting blood glucose at 2 weeks | 2 weeks
  After verifying fasting for 10-12 hours, a blood sample (about 15 ml, approximately 1 tablespoon) will be collected via venipuncture to measure markers of glucose. After withdrawal, blood will be centrifuged at 1,100 x g at 4°C for 20 minutes, and serum, plasma and erythrocytes will be aliquoted and stored at -80 degrees Celsius for subsequent analysis upon sample collection completion. Blood will be drawn by Arizona Biomedical Collaborative Laboratory clinical staff.
Change in femoral artery reactivity at 2 weeks | 2 weeks
  Femoral Artery Flow Mediated Dilation (FAFMD) Endothelium-dependent dilation of the femoral artery will be measured using B-mode ultrasound (Terason uSmart 3300+™, Burlington MA) using guidelines set forth by the Brachial Artery Reactivity Task Force.
Change in central aortic diastolic and systolic blood pressure at 2 weeks | 2 weeks
  All participants will lay down in a dimly lit room and have resting blood pressure measured using an automated blood pressure machine. Thereafter, an appropriately sized blood pressure cuff will be placed on the left arm and central and peripheral blood pressures will be assessed using the non-invasive SphygmoCor system.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilson SL, Crosley-Lyons R, Junk J, Hasanaj K, Larouche ML, Hollingshead K, Gu H, Whisner C, Sears DD, Buman MP. Effects of Increased Standing and Light-Intensity Physical Activity to Improve Postprandial Glucose in Sedentary Office Workers: Protocol for a Randomized Crossover Trial. JMIR Res Protoc. 2023 Aug 23;12:e45133. doi: 10.2196/45133. PMID 37610800